CLINICAL TRIAL: NCT04151004
Title: Functional Muscle Characteristics and Cardio-respiratory Interaction in Patients With Fontan Palliation
Acronym: FONTANEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FONTANEX_2019
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group (Experimental): Incremental cycling test to volitional exhaustion. Constant load cycling test to volitional exhaustion. Respiratory and leg muscle endurance test to volitional exhaustion. Three respiratory muscle training interventions.
  Interventions: Other: Incremental cycling test (ICT); Other: Constant load cycling test (CET); Other: Incremental respiratory muscle test (IncRMET); Other: Incremental quadriceps muscle test (IncQMT); Other: Respiratory muscle training like interventions
- Control group (Active Comparator): The control group executes the same tests as the patient group.
  Interventions: Other: Incremental cycling test (ICT); Other: Constant load cycling test (CET); Other: Incremental respiratory muscle test (IncRMET); Other: Incremental quadriceps muscle test (IncQMT); Other: Respiratory muscle training like interventions

INTERVENTIONS:
Other: Incremental cycling test (ICT) — Incremental cycling test to volitional exhaustion
Other: Constant load cycling test (CET) — Constant load cycling test to volitional exhaustion.
Other: Incremental respiratory muscle test (IncRMET) — Incremental respiratory muscle test to volitional exhaustion.
Other: Incremental quadriceps muscle test (IncQMT) — Incremental quadriceps muscle test to volitional exhaustion.
Other: Respiratory muscle training like interventions — Three different respiratory muscle training like interventions that are usually used for respiratory muscle trainings.

SUMMARY:
Congenital heart disease (CHD) is the most common congenital defect, affecting about 1% of newborns. Among adults surviving complex CHD, the cohort of survivors after the Fontan palliation for univentricular physiology is the most rapidly growing. Given their unique physiology without a pumping chamber supporting the pulmonary circulation, their exercise capacity as adults is often severely reduced. Therefore, patients with grown-up CHD typically need long-term expert medical care causing constantly increasing healthcare- related costs. Specific exercise regimes might offer a safe, efficacious and cost-effective alternative to pharmacologic interventions and surgery. The underlying mechanisms of impaired exercise capacity in Fontan patients are, however, not fully understood and consequently, training regimes specifically tackling the limiting factors cannot be developed. In patients with CHD, studies have suggested that exercise limitations are secondary to the cardiac defects, factors related to cardiac surgery, chronotropic incompetence and underlying lung disease. Similar to heart failure patients, exercise limitations could be traced back to insufficient respiratory and leg muscle functions and impaired cardiovascular regeneration processes possibly due to an altered stem cell number and function in the peripheral blood.

The present study will investigate cardiac, respiratory and quadriceps muscle function at rest and during submaximal and maximal whole-body exercises. A special focus will be given on respiratory and quadriceps muscle strength, and proneness of these muscles to fatigue, which has not yet been objectively investigated. Moreover, different respiratory muscle training (RMT) protocols will be executed, to assess the safety of these interventions. Moreover, the current study will be the first to investigate the influence of exhaustive exercise protocols on the number and function of circulating stem and progenitor cells (CPCs) in Fontan patients. The number of these cell populations was shown to strongly correlate with long-term outcome and recovery in several diseases. This study aims to reveal whether Fontan patients show similarly alternated stem cell number and function in the peripheral blood, that likely result in impaired vascular regeneration processes and possibly also contribute to reduced exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 55 years
* Fontan palliation (for Fontan patients)
* NYHA I - III (for Fontan patients)
* Willing to adhere to the study rules

Exclusion Criteria:

* NYHA IV (for Fontan patients)
* not being able to perform cycle exercise
* known diaphragmatic paresis
* being pregnant or breast feeding
* Intention to become pregnant during the course of the study
* known or suspected non-compliance, drug or alcohol abuse
* Regular intake of medication affecting sleep or the performance of the respiratory, cardiovascular or neuromuscular system (except for Fontan-related medication for patients)
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* previous enrolment in current study
* being investigator or his/her family member, employee or another dependent person

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change in respiratory muscle strength (in cmH2O) | At baseline and after acute exercise (approximately 15 minutes)
  Change in respiratory muscle strength will be measured between baseline and after an acute exercise
Change in quadriceps muscle strength (in Newton) | At baseline and after acute exercise (approximately 15 minutes)
  Change in quadriceps muscle strength will be measured between baseline and after an acute exercise

SECONDARY OUTCOMES:
Change in ventilation (in liter per minute) | On visit 1at baseline and after acute exercise (approximately 15 minutes)
  Change in ventilation will be measured between baseline and after an acute exercise
Change in gas exchange (in liter per minute) | At baseline and after acute exercise (approximately 15 minutes)
  Change in gas exchange will be measured between baseline and after an acute exercise
Change in heart rate (beats per minute) | At baseline and after acute exercise (approximately 15 minutes)
  Change in heart rate will be measured between baseline and after an acute exercise
Change in cardiac output (in liter per minute) | At baseline and after acute exercise (approximately 15 minutes)
  Change in cardiac output will be measured between baseline and after an acute exercise
Change in blood pressure (in mmHg) | At baseline and after acute exercise (approximately 15 minutes)
  Change in cardiac output will be measured between baseline and after an acute exercise
Change in blood oxygen saturation (in %) | At baseline and after acute exercise (approximately 15 minutes)
  Change in blood oxygen saturation will be measured between baseline and after an acute exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Physiology Lab, Institute of Human Movement Sciences and Sport, ETH Zurich, Zurich, Canton of Zurich, Switzerland